CLINICAL TRIAL: NCT04680741
Title: Application Based Addiction Treatment Adherence Trial: a Pilot Study
Brief Title: Application Based Addiction Treatment Adherence Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Open Health Network (Unknown)
Responsible Party: Principal Investigator, Robert Bales, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-636
Record Dates: First submitted 2020-09-03; First posted 2020-12-23 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2023-07

CONDITIONS: Opiate Use Disorder

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort pilot study to test the feasibility of a smartphone-based application (app) which is designed to monitor attendance at twelve-step facilitation meetings.
Masking Description: Primary Care provider (PI) will be blinded during the active enrollment and study phase of the trial. PI will continue to be the treating physician for these patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Addiction Pilot App (Experimental): Patients in this arm will be asked to use an application that works by allowing patients to check in to meetings and tracks patients' location for a period of 90 days.
  Patients will be asked to download the application to their smart phone. At each of patients' usual meetings we will ask patients to check in and check out of the meeting via the App. At the conclusion of this study patients may be invited to participate in a focus group.
  Interventions: Behavioral: Addiction Pilot App behavior tracking

INTERVENTIONS:
Behavioral: Addiction Pilot App behavior tracking — a smartphone-based application (app) which is designed to monitor attendance at twelve-step facilitation meetings.

SUMMARY:
The purpose of this study is to test a smart phone based application (the App) that will allow patients to record their attendance at 12-step meetings. The smart phone application is an investigational (experimental) application that works by allowing patients to check in to meetings and tracks their location. This application uses features available in smartphone technology and will be tested on a small scale in order to ascertain interest and benefit in a controlled manner. The initial phase of this process is a test of concept, which poses the question of whether individuals in an office-based addiction treatment program will utilize the application to check in and out of meetings, and answer a brief questionnaire delivered via the app at the end of a meeting. In this phase, investigators will set the standard recommendation as attendance at a minimum of three meetings per week.

DETAILED DESCRIPTION:
Treatment for addiction disorders has shown efficacy, but compliance with treatment is often a problem. Monitoring compliance in treatment is a difficult endeavor that is currently reliant on urine drug screens, monitoring of automated state pharmacy reporting systems, and requiring signature documentation of attendance at twelve-step meetings. These three methods are far from fool-proof and urine monitoring and signature documentation of meeting attendance are notoriously falsified by patients through a wide array of strategies. There is opportunity is to develop a smartphone application-based intervention protocol that will monitor individual's compliance with recommended attendance at prescribed twelve-step meetings. Investigators have partnered with Open Health Network to develop this application and currently have a working prototype.

Patients who are engaged in the twelve-step process have higher rates of continued sobriety as compared to patients who do not attend or are not engaged in the process. People with addiction have increased sobriety rates if they are accountable to someone outside of themselves. Therefore, investigators encourage patients to attend meetings frequently, have a sponsor, and actively work through the twelve steps. A sponsor is an individual who has been participating in a twelve-step facilitation program and has been sober for a minimum of one year. Leveraging technology to hold individuals accountable for participating in these meetings will improve their continued sobriety. A systematic review of available smartphone apps for alcohol and drug abuse, published in 2019, concluded that most did not incorporate evidence based addiction treatment. Furthermore, some apps promoted harmful drinking or substance abuse.

Investigators are interested in developing an application for mobile devices that will document 12-step meeting attendance in a way that is more reliable than the typical sign in sheet. This research study is a small trial that is designed to prove our concept and gather information for future development of the application.

Eligible patients will be asked to download the application to their smart phone. These patients will be asked to use the application for a period of 90 days. At each of patients' usual meetings investigators will ask patients to check in and check out of the meeting via the App. At the conclusion of this study patients may be invited to participate in a focus group.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, age 18 and over,
2. Currently being treated for opiate addiction at the family medicine clinic at the CCF South Pointe Campus.
3. Patients who have a smartphone (iOS or Android) or iPod Touch.
4. Patients who are engaged with a twelve-step program.

Exclusion Criteria:

1. Patients who are not willing to install the application to their personal phone.
2. Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
meeting attendance frequency | from baseline to up to 90 days
  collected via the participant's smart phone
sponsor contact frequency | from baseline to up to 90 days
  collected via the participant's smart phone
feedback and ecological mental and physical health assessment | from baseline to up to 90 days
  collected via the participant's smart phone after each meeting attendance. An item asking whether or not the meeting was helpful (yes / no). 7-item simplified ecological assessment designed for a 10-second snapshot of patients' mental and physical health status. It is visual analog scale of 0 to 10 on Mood (very poor - excellent), anxiety (very anxious - calm), stress (very stressed - relaxed), sleep (insomnia - full night), decision making (Brain fog - clarity), exercise (None - >90 minutes). The scale was developed by Open Health Network investigator and has not been validated. Each score will be tracked for changes over time but there won't be composite scores.
clinical markers of sobriety (1) | most recent test results from baseline to up to 90 days (+/- 30 days)
  Urine will be screened for the presence/absence of the following substances:
  1. Cannabinoid
  2. Benzylecognine
  3. 6-Acetylmorphine
  4. Amphetamine
  5. Methamphetamine
  6. Buprenorphine
  7. Norbuprenorphine
  8. Methadone
  9. EDDP
  10. Tramadol
  11. Desmethyltramadol
  12. Fentanyl
  13. Norfentanyl
  14. Codeine
  15. Morphine
  16. Dihydrocodeine
  17. Hydrocodone
  18. Oxycodone
  19. Hydromorphone
  20. Oxymorphone
clinical markers of sobriety (2) | most recent test results from baseline to up to 90 days (+/- 30 days)
  Urine will be screened for value changes in the following:
  21. Urine pH (date and result) 22. Specific gravity
clinical markers of sobriety (3) | most recent test results from baseline to up to 90 days (+/- 30 days)
  Urine will be screened for the presence/absence of the following substances:
  23. Oxidants 24. Nitrites 25. Chromate
clinical markers of sobriety (4) | most recent test results from baseline to up to 90 days (+/- 30 days)
  Urine will be screened for the presence/absence of the following substances:
  Phencyclidine Benzodiazepines Cocaine Opiates Barbiturates Ethanol
Treatment visit frequency | from baseline to up to 90 days
  treatment dates (visit frequency) will be extracted from Electric Health Record(EHR)
Treatment dose changes | from baseline to up to 90 days
  Buprenorphine (Suboxone, Subutex, Zubsolv, Bunavail) treatment dose changes will be tracked via EHR

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bales, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic South Pointe Hospital, Warrensville Heights, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1) Massatti, R., Beeghly C., Hall, O., Kariisa, M. & Potts, L. (2014, April). Increasing Heroin Overdoses in Ohio: Understanding the Issue. Columbus, OH: Ohio Department of Mental Health and Addiction Services.
- [Background] Laudet AB. The impact of alcoholics anonymous on other substance abuse-related twelve-step programs. Recent Dev Alcohol. 2008;18:71-89. doi: 10.1007/978-0-387-77725-2_5. PMID 19115764
- [Background] http://med.ohio.gov/LawsRules/NewlyAdoptedandProposedRules.aspx. 4731-11-12: Office based opioid treatment
- [Background] Ostling PS, Davidson KS, Anyama BO, Helander EM, Wyche MQ, Kaye AD. America's Opioid Epidemic: a Comprehensive Review and Look into the Rising Crisis. Curr Pain Headache Rep. 2018 Apr 4;22(5):32. doi: 10.1007/s11916-018-0685-5. PMID 29619569
- [Background] American Psychiatric Association, Diagnostic and Statistical Manual of Mental Disorders, fifth edition, 2013. ISBN: 978-0-89042-555-8
- [Background] Edelman EJ, Oldfield BJ, Tetrault JM. Office-Based Addiction Treatment in Primary Care: Approaches That Work. Med Clin North Am. 2018 Jul;102(4):635-652. doi: 10.1016/j.mcna.2018.02.007. PMID 29933820
- [Background] Nissly T, Levy R. Buprenorphine to treat opioid use disorder: A practical guide. J Fam Pract. 2018 Jun;67(9):544-548. PMID 30216393
- [Background] US Department of Health and Human Services/Centers for Disease Control and Prevention. MMWR / January 4, 2019 / Vol. 67 / Nos. 51 & 52
- [Background] Tofighi B, Chemi C, Ruiz-Valcarcel J, Hein P, Hu L. Smartphone Apps Targeting Alcohol and Illicit Substance Use: Systematic Search in in Commercial App Stores and Critical Content Analysis. JMIR Mhealth Uhealth. 2019 Apr 22;7(4):e11831. doi: 10.2196/11831. PMID 31008713